CLINICAL TRIAL: NCT04070846
Title: A Phase 1, Open-Label, Single-Dose, Mass Balance Study to Evaluate the Absorption, Metabolism, and Excretion of [14C]-LC350189 in Healthy Male Subjects
Brief Title: Mass Balance Study of [14C]LC350189 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LG-GDCL005
Record Dates: First submitted 2019-08-19; First posted 2019-08-28 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C] LC350189 (Experimental): Single oral dose
  Interventions: Drug: [14C] LC350189

INTERVENTIONS:
Drug: [14C] LC350189 — Carbon-14 labelded LC350189

SUMMARY:
This is a Phase 1, open-label, single-dose, mass balance study designed to evaluate the absorption, metabolism, and excretion of [14C] radiolabeled LC350189 after oral administration.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male 18 to 55 years of age, inclusive.
* The subject has a body mass index 18 to 32 kg/m2, inclusive, at screening.
* The subject is judged by the investigator to be in good general health, as determined by medical history, clinical laboratory assessments, vital sign measurements, 12 lead electrocardiogram results, and physical examination findings at screening.
* The subject is able to provide written informed consent.

Exclusion Criteria:

* The subject has a medical history of any issues affecting absorption or metabolism, as judged by the investigator.
* The subject has a medical history of any problems affecting venous access or bowel/bladder function.
* The subject has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies at screening.
* The subject has used any prescription or over the counter medications (except paracetamol [up to 2 g per day]), including herbal or nutritional supplements, within 14 days before the first dose of study drug.
* The subject has consumed grapefruit or grapefruit juice, Seville orange or Seville orange containing products (eg, marmalade), or caffeine- or xanthine containing products within 48 hours before the first dose of study drug or during the study.
* The subject has a positive test result for drugs of abuse, alcohol, or cotinine (indicating active current smoking) at screening or before the first dose of study drug.
* The subject is involved in strenuous activity or contact sports within 24 hours before the first dose of study drug or during the study.
* The subject has donated blood or blood products >450 mL within 30 days before the first dose of study drug.
* The subject has a history of relevant drug and/or food allergies (ie, allergy to study drug or excipients, or any significant food allergy that could preclude a standard diet in the clinical unit).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2020-03-07 (Actual); Study Completion 2020-03-07 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery of total radioactivity in whole blood and plasma. | Before dosing on Days 1 through Day 10 (240 hours)
  Radioactivity is measured by radiation dosimetry.
Mass balance recovery of total radioactivity in whole urine, and feces. | Before dosing on Days 1 through Day 10 (240 hours)
  Radioactivity is measured by radiation dosimetry.

SECONDARY OUTCOMES:
Incidence of adverse events | form baseline up to Day 11
  Safety

CONTACTS AND LOCATIONS:
Locations (1):
- PPD, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided